CLINICAL TRIAL: NCT02187926
Title: Observational Study for the Evaluation of Clinical Effectiveness in Routine Practice of Daxas® (Roflumilast), in Approximately 2700 Patients With Severe and Very Severe COPD (Chronic Obstructive Pulmonary Disease) in Greece
Brief Title: Evaluation of Clinical Effectiveness of Roflumilast in Routine Practice, in Chronic Obstructive Pulmonary Disease (COPD) Patients in Greece
Acronym: ATLAS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: RO-2455-401-GR
Record Dates: First submitted 2014-04-29; First posted 2014-07-11 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Drug therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Roflumilast: Roflumilast will be administered according to the prescribing information of the approved label in Greece.

SUMMARY:
The purpose of this study was to examine the characteristics of patients selected for treatment with roflumilast and the effectiveness and safety of roflumilast in patients with severe or very severe COPD treated in Hospital and outpatient specialist ward settings in Greece.

DETAILED DESCRIPTION:
The drug being observed in this study is called roflumilast. Roflumilast is used to treat people who have chronic obstructive pulmonary disease (COPD) associated with chronic bronchitis with a history of worsening symptoms. This study looked at side effects and the lung function of people who take roflumilast. The study enrolled 2577 patients who were already prescribed roflumilast as an add on to bronchiodilator treatment by their healthcare provider. This multi-centre trial was conducted in Greece. The overall time to participate in this study was up to 6 months. Participants were evaluated during routine appointments with their healthcare provider.

ELIGIBILITY:
Inclusion Criteria

* Be diagnosed with COPD at stages 3 or 4 according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines.
* Have the clinical phenotype of chronic bronchitis with cough and sputum production (with or without emphysema).
* Already be receiving treatment for their disease (inhaled bronchodilators (long-acting beta2-agonists (LABA), long-acting muscarinic antagonists (LAMA), short-acting beta2-agonists (SABA), short-acting muscarinic antagonist (SAMA)), inhaled corticosteroids (ICS), combination of inhaled bronchodilators and corticosteroids.
* Be aged over 40 years

Exclusion Criteria:

• None

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients prescribed roflumilast in Greece.
Sampling Method: Non-Probability Sample
Enrollment: 2577 (Actual)
Dates: Start 2011-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Forced Expiratory Volume in First Second (FEV1) at Month 6 | Baseline and Month 6
  FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation.
Change From Baseline in Forced Vital Capacity (FVC) at Month 6 | Baseline and Month 6
  Vital capacity is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible.
Change From Baseline in Ratio of Forced Expiratory Volume After 1 Second to Forced Vital Capacity (FEV1/FVC) at Month 6 | Baseline and Month 6
  The FEV1/FVC ratio represents the percentage of vital capacity expelled from the lungs during the first second of a forced exhalation.

SECONDARY OUTCOMES:
Change from Baseline in Forced Expiratory Volume in First Second (FEV1) at Month 6 | Baseline and Month 6
  FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation.
Percentage of Participants with Chronic Obstructive Pulmonary Disease (COPD) Exacerbations | Month 3 and Month 6
  A COPD exacerbation is an event characterised by a worsening in the patient's baseline dyspnoea, or cough and/or sputum beyond day-to-day variability sufficient to warrant a change in management, and may be accompanied by increased wheeze, chest tightness, purulent sputum and symptoms of cold and/or fatigue.
Percentage of Participants requiring Hospitalizations due to Exacerbations of COPD | Up to Month 6
Change from Baseline in Clinical COPD Questionnaire (CCQ) Total Score | Baseline and Months 3 and 6
  Quality of life will be evaluated using the Clinical COPD Questionnaire (CCQ) 10-item questionnaire. The questions in the CCQ are divided into three area's, or domains: Symptoms: items 1, 2, 5 and 6; Functional state: items 7, 8, 9 and 10; Mental state: items 3 and 4. Individual items within the CCQ are equally weighted. The total score is calculated by adding the scores of the ten items and dividing that number by ten (= number of items). The total CCQ score, and the score on each of the three domains, varies between 0 (very good health status) to 6 (extremely poor health status).
Change from Baseline in MRC Dyspnea Scale | Baseline and Months 3 and 6
  The Medical Research Council (MRC) breathlessness (dyspnea) scale comprises five statements that describe almost the entire range of respiratory disability: 1 - Not troubled by breathlessness except on strenuous exercise; 2 - Short of breath when hurrying or walking up a slight hill; 3 - Walks slower than contemporaries on level ground because of breathlessness, or has to stop for breath when walking at own pace; 4 - Stops for breath after walking about 100m or after a few minutes on level ground; 5 - Too breathless to leave the house, or breathless when dressing or undressing. The highest numbered question to which the subject answered 'Yes' is the Dyspnea Scale Score.
Patient's Satisfaction with Roflumilast | Baseline and Months 3 and 6
  Is the perception of the participant according to the scale provided.
Physician's Satisfaction with Roflumilast | Baseline and Months 3 and 6
  Is the perception of Physician taking into consideration the effectiveness and the tolerability of the drug.
Change From Baseline in Forced Vital Capacity (FVC) at Month 3 | Baseline and Month 3
  Vital capacity is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible.
Change From Baseline in Ratio of Forced Expiratory Volume After 1 Second to Forced Vital Capacity (FEV1/FVC) at Month 3 | Baseline and Month 3
  The FEV1/FVC ratio represents the percentage of vital capacity expelled from the lungs during the first second of a forced exhalation.
Compliance to treatment | 6 months
  According to physician's judgment
Number of participants with adverse drug reactions (ADR) | 6 months
  An ADR is any response to a medicinal product which is noxious and unintended and which occurs at doses normally used in man for the prophylaxis, diagnosis or therapy of diseases or for the restoration, correction or modification of physiological function.
Concomitant administration of inhaled bronchodilators and corticosteroids | 6 months
  Concomitant administration of inhaled bronchodilators and corticosteroids, either separately or in combination.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca